CLINICAL TRIAL: NCT03417687
Title: Evaluation of Hyperpolarized 129Xe MRI as Compared to 133Xe Scintigraphy for the Assessment of Pulmonary Function in Patients Being Evaluated for Possible Lung Resection Surgery
Brief Title: Hyperpolarized Xenon MRI for Assessment of Pulmonary Function in Lung Resection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Polarean, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: POL-Xe-001
Record Dates: First submitted 2018-01-25; First posted 2018-01-31 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Pulmonary Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Open label crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): Subjects will undergo hyperpolarized 129Xe MRI first, followed by 133Xe scintigraphy
  Interventions: Drug: 129Xe MRI; Drug: 133 Xe scintigraphy
- Arm 2 (Active Comparator): Subjects will undergo 133Xe scintigraphy first, followed by hyperpolarized 129Xe MRI
  Interventions: Drug: 129Xe MRI; Drug: 133 Xe scintigraphy

INTERVENTIONS:
Drug: 129Xe MRI — Evaluation of pulmonary function
  Other Names: 129Xenon scintigraphy
Drug: 133 Xe scintigraphy — Evaluation of pulmonary function
  Other Names: 133Xenon scintigraphy

SUMMARY:
This study compares the equivalence of hyperpolarized 129Xe MRI as compared to 133Xe scintigraphy for the evaluation of pulmonary function in patients being evaluated for lung resection.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, cross-over Phase 3 study evaluating hyperpolarized 129Xe gas MRI as compared to 133Xe scintigraphy for the evaluation of pulmonary function. This study will enroll subjects being evaluated for possible lung resection surgery (i.e. segmentectomy, lobectomy, or pneumonectomy). Subjects will have both a 129Xe MRI and 133Xe scintigraphy image. The vast differences in technique for obtaining hyperpolarized 129Xe MRI as compared to 133Xe scintigraphy make it impossible to blind study procedures. However, all image interpretation will be performed by personnel blinded to the subject's medical history and all study assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 years of age.
2. Subject is being evaluated for possible lung resection (e.g., segmentectomy, lobectomy, or pneumonectomy).
3. Subject is able to undergo MRI imaging and able to fit in the MRI coil.
4. Subject is willing and able to comply with all study procedures.
5. Subject must understand and voluntarily sign an informed consent form (ICF) prior to any study specific assessments or procedures.

Exclusion Criteria:

1. Baseline blood oxygen saturation (SpO2) <90% at rest. For patients requiring routine supplemental oxygen, SpO2 measurements should be taken with the patient's normal oxygen supplementation.
2. Female subjects of childbearing potential with a positive serum pregnancy test at screening, or who are not taking (or not willing to take) acceptable birth control measures through the Follow-up Period. Adequate birth control methods include with a monogamous partner who was sterilized more than 6 months prior to screening, or measures with a Pearl index of <1 used consistently and correctly (including intrauterine devices, or implantable, injectable, oral, or transdermal contraceptives). Women are not considered to be of childbearing potential if they meet at least 1 of the following 2 criteria as documented by the Investigator:

   * They have had a hysterectomy, bilateral salpingectomy, or bilateral oophorectomy at a minimum of 1 menstrual cycle prior to signing the ICF; or
   * They are post-menopausal: for women ≥55 years of age, defined as ≥1 year since their last menstrual period, or for women <55 years of age, defined as ≥1 year since their last menstrual period and have a follicle-stimulating hormone (FSH) level in the laboratory's normal range for post-menopausal phase.
3. Women who are lactating and insist on breast feeding.
4. Subjects who have received any other investigational therapy within 4 weeks prior to Screening.
5. Subjects who require anesthesia or heavy sedation to undergo MRI testing. Mild sedation could be acceptable (i.e. a low dose oral acting anxiolytic medication such as alprazolam) as long as, in the opinion of the investigator, the subject meets Inclusion Criteria #4 and #5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth P West, Study Director — Polarean, Inc.
Locations (3):
- United States (3):
  - Duke University Hospital, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 129Xe Before 133Xe: Subjects will undergo hyperpolarized 129Xe MRI first, followed by 133Xe scintigraphy
  129Xe MRI: Evaluation of pulmonary function
  133 Xe scintigraphy: Evaluation of pulmonary function
- 133Xe Before 129Xe: Subjects will undergo 133Xe scintigraphy first, followed by hyperpolarized 129Xe MRI
  129Xe MRI: Evaluation of pulmonary function
  133 Xe scintigraphy: Evaluation of pulmonary function
Period: Overall Study
Arm/Group | 129Xe Before 133Xe | 133Xe Before 129Xe
Started | 18 (4 subjects were randomized to the 129Xe before 133Xe group but discontinued prior to receiving the first treatment.) | 20
Received 129Xe | 14 | 20
Received 133Xe | 13 | 20
Completed | 14 | 20
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Population: Number of baseline participants is based on the safety analysis set. The safety analysis set includes all subjects that received at least 1 dose of study drug. 4 randomized subjects in the 129Xe before 133Xe group discontinued prior to receiving any dose of study drug and thus were not included in the safety analysis set.
Groups:
- Total: Total of all reporting groups
Arm/Group | 129Xe Before 133Xe | 133Xe Before 129Xe | Total
Number analyzed (Participants) | 14 | 20 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (11.5) | 64.9 (7.6) | 62.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 9 | 14 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 20 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 12 | 15 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 20 | 34

OUTCOME MEASURES:

1. Primary Outcome: Predicted Percentage of Remaining Pulmonary Function
Description: Predicted percentage of remaining pulmonary function is a pre-specified section of lung were to be removed. Investigators indicated which portions of lung were likely to be resected. Remaining percentage of pulmonary function was determined by subtracting the percentage of pulmonary function contributed by the planned zone of resection from the total pulmonary function using a standard 6-zone image analysis of the lung. The difference between predicted percentage of remaining pulmonary function was calculated by subtracting the value derived from the 133Xe scintigraphy image from the value derived from the 129Xe MRI image (e.g. 129Xe - 133Xe).
Time Frame: 48 hours
Population: The Efficacy Analysis Set is the group of subjects who had both a 129Xe MRI scan and a 133Xe scintigraphy scan, and for whom both scans met quality control criteria for analysis (as defined in the Independent Review Charter).
Measure: Mean (Standard Deviation); unit: percentage of remaining function
Groups:
- 129Xe MRI: All subjects receiving a 129Xe MRI of their lungs. Subjects received both 129Xe MRI and 133Xe scintigraphy in randomized order.
- 133Xe: All subjects receiving a 133Xe scintigraphy scan of their lungs. Subjects received both 129Xe MRI and 133Xe scintigraphy in randomized order.
Arm/Group | 129Xe MRI | 133Xe
Number analyzed (Participants) | 32 | 32
percentage of remaining function | 73.4 (13.0) | 71.9 (12.1)
Statistical Analysis 1: Comparison: 129Xe MRI vs 133Xe; The primary efficacy analysis tested the mean difference in the predicted percentage of remaining pulmonary function as measured by 129Xe MRI relative to the value as measured by 133Xe scintigraphy (reference standard) if a pre-defined section of lung were resected; Test type: Equivalence — The 2 methods were considered equivalent if the 95% confidence interval for the mean within subject difference between 129Xe MRI and 133Xe scintigraphy measurements was contained within the equivalence margin (-14.7%, +14.7%); Mean Difference (Net) = 1.4, 95% CI 2-sided [-0.75 to 3.60], Standard Deviation 5.9

2. Secondary Outcome: Predicted Versus Measured FEV1
Description: The difference between the scan-predicted post-operative FEV1 and the measured post-operative FEV1
Time Frame: 3 months
Population: This analysis set of all subjects that met the criteria for inclusion in the efficacy analysis set and had a post-operative FEV1 (spirometry) value.
Measure: Mean (Standard Deviation); unit: liters
Groups:
- 129Xe MRI: Subjects receiving 129Xe MRI. All subjects received 129Xe MRI and 133Xe scintigraphy in randomized order.
- 133Xe Scintigraphy: Subjects receiving 133Xe scintigraphy. All subjects received 129Xe MRI and 133Xe scintigraphy in randomized order.
Arm/Group | 129Xe MRI | 133Xe Scintigraphy
Number analyzed (Participants) | 32 | 32
liters | -0.65 (0.60) | -0.65 (0.66)

3. Secondary Outcome: Measured Percentage of Total Ventilation Contributed by the Lower Left Lung Zone.
Description: The fraction of total ventilation contributed by the lower left lung zone on 6-zone analysis.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: percentage of total function
Groups:
- 129Xe MRI: All subjects receiving 129Xe MRI. Subjects received both 129Xe MRI and 133Xe scintigraphy in randomized order.
- 133Xe Scintigraphy: All subjects receiving 133Xe scintigraphy. Subjects received both 129Xe MRI and 133Xe scintigraphy in randomized order.
Arm/Group | 129Xe MRI | 133Xe Scintigraphy
Number analyzed (Participants) | 32 | 32
percentage of total function | 16.08 (4.43) | 12.37 (3.60)
Statistical Analysis 1: Comparison: 129Xe MRI vs 133Xe Scintigraphy; Test type: Equivalence — The 2 methods were considered equivalent if the 95% confidence interval for the mean within subject difference between 129Xe MRI and 133Xe scintigraphy measurements was contained within the equivalence margin (-5.0%, +5.0%); Mean Difference (Final Values) = 3.71, 95% CI 2-sided [2.12 to 5.29], Standard Deviation 4.39

4. Secondary Outcome: Measured Percentage of Total Ventilation Contributed by the Upper Left Lung Zone.
Description: The fraction of total ventilation contributed by the upper left lung zone on 6-zone analysis.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: percentage of total function
Groups:
- 129Xe MRI: Subjects receiving 129Xe MRI. All subjects received 129Xe MRI and 133 Xe scintigraphy in randomized order.
- 133Xe Scintigraphy: Subjects receiving 133Xe scintigraphy. All subjects received 129Xe MRI and 133 Xe scintigraphy in randomized order.
Arm/Group | 129Xe MRI | 133Xe Scintigraphy
Number analyzed (Participants) | 32 | 32
percentage of total function | 10.67 (2.11) | 10.28 (2.72)
Statistical Analysis 1: Comparison: 129Xe MRI vs 133Xe Scintigraphy; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.390, 95% CI 2-sided [-0.476 to 1.26], Standard Deviation 2.40

5. Secondary Outcome: Measured Percentage of Total Ventilation Contributed by the Middle Left Lung Zone.
Description: The fraction of total ventilation contributed by the middle left lung zone on 6-zone analysis.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: percentage of total function
Arm/Group | 129Xe MRI | Arm 2
Number analyzed (Participants) | 32 | 32
percentage of total function | 22.27 (3.71) | 20.92 (2.88)
Statistical Analysis 1: Comparison: 129Xe MRI vs Arm 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 1.35, 95% CI 2-sided [0.184 to 2.505], Standard Deviation 3.22

6. Secondary Outcome: Measured Percentage of Total Ventilation Contributed by the Upper Right Lung Zone.
Description: The fraction of total ventilation contributed by the upper right lung zone on 6-zone analysis.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: percentage of total function
Arm/Group | 129Xe MRI | 133Xe Scintigraphy
Number analyzed (Participants) | 32 | 32
percentage of total function | 11.16 (2.97) | 12.12 (2.56)
Statistical Analysis 1: Comparison: 129Xe MRI vs 133Xe Scintigraphy; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-2.101 to 0.181], Standard Deviation 3.16

7. Secondary Outcome: Measured Percentage of Total Ventilation Contributed by the Middle Right Lung Zone.
Description: The fraction of total ventilation contributed by the middle right lung zone on 6-zone analysis.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: percentage of total function
Groups:
- 133 Xe Scintigraphy: Subjects receiving 133Xe scintigraphy. All subjects received 129Xe MRI and 133Xe scintigraphy in randomized order.
Arm/Group | 129Xe MRI | 133 Xe Scintigraphy
Number analyzed (Participants) | 32 | 32
percentage of total function | 23.44 (3.07) | 26.16 (3.80)
Statistical Analysis 1: Comparison: 129Xe MRI vs 133 Xe Scintigraphy; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -2.721, 95% CI 2-sided [-4.096 to -1.345], Standard Deviation 3.82

8. Secondary Outcome: Measured Percentage of Total Ventilation Contributed by the Lower Right Lung Zone.
Description: The fraction of total ventilation contributed by the lower right lung zone on 6-zone analysis.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: percentage of total function
Arm/Group | 129Xe MRI | 133Xe Scintigraphy
Number analyzed (Participants) | 32 | 32
percentage of total function | 16.39 (4.18) | 18.16 (3.62)
Statistical Analysis 1: Comparison: 129Xe MRI vs 133Xe Scintigraphy; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.76, 95% CI 2-sided [-3.192 to -0.335], Standard Deviation 3.96

ADVERSE EVENTS:
Time Frame: 3 days
Description: All subjects were dosed with 129Xe and 133Xe on the same day with a mean time between administration of 1.8 hours (range 0.7 hours to 4.9 hours). Therefore reported adverse events could not reliably be attributed to an individual drug. Therefore, adverse events are reported based on the randomized order to which participants received each drug.
Arm/Group | 129Xe Before 133Xe | 133Xe Before 129Xe
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/20
Other Adverse Events (participants affected / at risk) | 2/14 | 3/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 129Xe Before 133Xe (N=14) | 133Xe Before 129Xe (N=20)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 129Xe Before 133Xe (N=14) | 133Xe Before 129Xe (N=20)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hair disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Independent analyses and/or publication of trial results by the PI is not permitted without prior written consent of the sponsor. Written permission to investigators to publish results is contingent on review by the sponsor of the methodology and statistical analyses used. The PI must submit all manuscripts to the sponsor at least 60 days prior to submission for review.

DOCUMENTS (2):
  • Study Protocol (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/87/NCT03417687/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT03417687/SAP_001.pdf